CLINICAL TRIAL: NCT05539677
Title: Analysis of the Immunogenetic Profile of Patients With Aggressive Course of Malignant Neoplastic Process Resistant to the Standard Treatment Approaches: a Translational Study
Brief Title: Biobank and Register of Patients With Agresive Tumors for Translational and Analytical Research
Acronym: REGATA
Status: Recruiting | Type: Observational
Sponsor: N.N. Petrov National Medical Research Center of Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: AAAA-A18-118032890188-9
Record Dates: First submitted 2022-09-04; First posted 2022-09-14 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Malignant Solid Tumors; Primary Brain Tumor; Melanoma; Soft Tissue Sarcoma; Colorectal Cancer; Kidney Cancer; Prostate Cancer
MeSH Terms: conditions — Brain Neoplasms; Melanoma; Sarcoma; Colorectal Neoplasms; Kidney Neoplasms; Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Blood, peripheral blood mononuclear cells, plasma, serum, living tumor tissue, archive tumor tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Melanoma
- Soft tissue sarcoma
- Kidney cancer
- Primary brain tumors
- Malignant neoplasms
- Prostate cancer
- Colorectal cancer

SUMMARY:
The investigators will collect biosamples of patient blood and tumour tissue for further immunological analysis of blood cell subpopulations, immunosupressive factors concentration, HLA expression an lymphocytes and tumour tissue, and and cancer testis antigenes expression on tumour cells, as well as clinical data on patient's stage, therapy, response and demographics. Possible prognostic and predictive dynamic biomarkers will be discovered for individualisation of treatment strategies

ELIGIBILITY:
Inclusion Criteria:

* Signed inform consent
* Histolgically verified solid tumour
* Receiving systemic therapy for neoplasm
* Has archival tumour tissue
* Provide biosamples with living tumour tissue or blood samples for immunologic assessment

Exclusion Criteria:

* Concurrent Lymphoprolipherative disorder
* Patients after stem cell or bone marrow thansplantation
* Incomplete informaton on previous cancer history or medical history
* Patients with known primary immunodeficiency
* Patients receiving immunosupressive therapy for concurrent illness
* Pregnant patients

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will include patients with solid tumours receiving systemic therapy for their disease who do not have other significant factors that affect the immune system
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 1998-09 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Progression in 3 mo | 3 month
  Presence of disease progression within 3 mo from sample aquisition

SECONDARY OUTCOMES:
Overall survival (OS) | Up to 5 years
  Time from sample aquisition to death from any reason
Progression free survival | Up to 5 years
  Time from sample aquisition to progression or death from the disease
Response rate | During the intervention
  Response assesmenr with RECIST 1.1 and iRECIST

CONTACTS AND LOCATIONS:
Overall Officials: Irina Baldueva, MD, PhD, DSc, Study Director — N.N. Petrov NMRC of Oncology
Locations (1):
- N.N. Petrov NMRC of Oncology, Oncoimmunology dep., Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: Undecided
Upon completion, the database is planned to be published with depersonalized data for cohorts with meaningful data. Cohorts to be published will be defined upon data check. Partial publications could be applicable.

REFERENCES:
- [Result] Shendaleva N, Novik AV, Zozulya A, Nekhaeva TL, Semenova A, Teletaeva GM, et al. Impact of the azoximer bromide concomitant therapy on patient outcomes in patients with melanoma. Journal of clinical oncology : official journal of the American Society of Clinical Oncology. 2021;39(15_suppl):e21574-e.
- [Result] Novik AV, Shendaleva N, Zozulya A, Nekhaeva TL, Semenova A, Teletaeva GM, et al. Impact of the azoximer bromide concomitant therapy on outcomes in patients with soft tissue sarcoma. Journal of clinical oncology : official journal of the American Society of Clinical Oncology. 2021;39(15_suppl):e23534-e.
- [Result] Novik AV, Girdyuk DV, Nekhaeva TL, Emelyanova NV, Semenova A, Teletaeva GM, et al. Progression prediction model for solid tumors with clinical and immunological parameters. Journal of clinical oncology : official journal of the American Society of Clinical Oncology. 2021;39(15_suppl):2539.